CLINICAL TRIAL: NCT06916676
Title: Optimal High-Intensity Laser Therapy (HILT) Parameters for Pain and Function in Patients With Moderate Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: HILT Dose Optimization for Knee Osteoarthritis Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al Hayah University In Cairo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HILT-KOA-DOSE
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low-Dose HILT (10 J/cm²) (Experimental): Participants receive High-Intensity Laser Therapy at a dosage of 10 J/cm² per treatment zone, 3 times per week for 4 weeks (12 sessions total).
  Interventions: Device: Low-Dose High-Intensity Laser Therapy (10 J/cm²)
- Medium-Dose HILT (15 J/cm²) (Experimental): Participants receive High-Intensity Laser Therapy at a dosage of 15 J/cm² per treatment zone, 3 times per week for 4 weeks (12 sessions total).
  Interventions: Device: Medium-Dose High-Intensity Laser Therapy (15 J/cm²)
- High-Dose HILT (20 J/cm²) (Experimental): Participants receive High-Intensity Laser Therapy at a dosage of 20 J/cm² per treatment zone, 3 times per week for 4 weeks (12 sessions total).
  Interventions: Device: High-Dose High-Intensity Laser Therapy (20 J/cm²)
- Sham HILT (Sham Comparator): Participants receive a sham High-Intensity Laser Therapy procedure using the same device and application technique, but with no energy delivered, 3 times per week for 4 weeks (12 sessions total).
  Interventions: Device: Sham High-Intensity Laser Therapy

INTERVENTIONS:
Device: Low-Dose High-Intensity Laser Therapy (10 J/cm²) — Application of HILT using an Nd:YAG laser (BTL-6000, 1064 nm). Delivered via continuous scanning technique (1 cm distance) to 5 zones (25 cm² each) covering anterior, medial, and lateral knee aspects. Target dose: 10 J/cm² per zone. Session frequency: 3x/week for 4 weeks (12 total). Session duration: 15-20 min. Administered by trained PTs in outpatient rehab. Skin temperature monitored.
  Arms: Low-Dose HILT (10 J/cm²)
Device: Medium-Dose High-Intensity Laser Therapy (15 J/cm²) — Application of HILT using an Nd:YAG laser (BTL-6000, 1064 nm). Delivered via continuous scanning technique (1 cm distance) to 5 zones (25 cm² each) covering anterior, medial, and lateral knee aspects. Target dose: 15 J/cm² per zone. Session frequency: 3x/week for 4 weeks (12 total). Session duration: 15-20 min. Administered by trained PTs in outpatient rehab. Skin temperature monitored.
  Arms: Medium-Dose HILT (15 J/cm²)
Device: High-Dose High-Intensity Laser Therapy (20 J/cm²) — Application of HILT using an Nd:YAG laser (BTL-6000, 1064 nm). Delivered via continuous scanning technique (1 cm distance) to 5 zones (25 cm² each) covering anterior, medial, and lateral knee aspects. Target dose: 20 J/cm² per zone. Session frequency: 3x/week for 4 weeks (12 total). Session duration: 15-20 min. Administered by trained PTs in outpatient rehab. Skin temperature monitored.
  Arms: High-Dose HILT (20 J/cm²)
Device: Sham High-Intensity Laser Therapy — Sham procedure mimicking active HILT using the same Nd:YAG laser device (BTL-6000). Same setup, patient positioning, scanning technique over identical zones, and session duration/frequency (3x/week, 4 weeks, 15-20 min). Device powered on with visual/auditory cues active, but no laser energy emitted. Administered by trained PTs in outpatient rehab. Skin temperature monitored.
  Arms: Sham HILT

SUMMARY:
This study aims to find the best settings (dose) for High-Intensity Laser Therapy (HILT) to reduce pain and improve function in people with moderate knee osteoarthritis. Participants will be randomly assigned to receive one of three different doses of HILT (low, medium, or high) or a sham (placebo) laser treatment, three times a week for four weeks. The main outcomes measured will be changes in knee pain (using a pain scale) and knee function (using a questionnaire) from the beginning to the end of the 4-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

Age between 45 and 75 years, inclusive. Clinical diagnosis of knee osteoarthritis according to American College of Rheumatology (ACR) criteria (knee pain plus at least 3 of 6: age >50, morning stiffness <30 min, crepitus, bony tenderness, bony enlargement, no palpable warmth).

Radiographic evidence of knee osteoarthritis corresponding to Kellgren-Lawrence grade II or III in the target knee.

Average knee pain intensity ≥ 4 on a 10-cm Visual Analogue Scale (VAS) during weight-bearing activities in the past week.

Willingness and ability to attend 3 sessions per week for 4 weeks and attend all assessment sessions.

Exclusion Criteria:

Previous surgery on the index knee (including arthroscopy within the last year or joint replacement).

Diagnosis of inflammatory arthritis (e.g., rheumatoid arthritis, psoriatic arthritis, gout).

Intra-articular corticosteroid or hyaluronic acid injection in the index knee within the last 3 months.

Clinically significant comorbidities that could interfere with participation or assessment (e.g., severe uncontrolled cardiovascular disease, severe pulmonary disease, significant neurological deficits affecting the lower limb).

Presence of skin conditions (e.g., infection, open wounds, eczema, photosensitivity disorders) in the area designated for laser treatment.

Current use of anticoagulant medication (e.g., warfarin, DOACs) due to potential risk, unless stable and cleared by physician. (Consider if this is truly necessary based on HILT mechanism).

History of cancer in the treatment area or active malignancy elsewhere. Known photosensitivity or use of photosensitizing medications. Pregnancy, planning pregnancy, or breastfeeding. Participation in another interventional clinical trial within the last 30 days. Inability to understand or communicate in the study language.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-04-23 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Pain Intensity | Baseline (T0), Mid-treatment (T1 - after 6 sessions), Post-treatment (T2 - after 12 sessions), 3-month Follow-up (T3)
  Visual Analogue Scale (VAS) for Pain: Change from baseline in average knee pain over the past week, measured on a 10 cm horizontal VAS, where 0 cm = no pain and 10 cm = worst imaginable pain. Higher scores indicate worse pain. Minimal Clinically Important Difference (MCID) estimated at 1.25 cm.
Change in Knee Osteoarthritis Symptoms and Function | Baseline (T0), Mid-treatment (T1), Post-treatment (T2), 3-month Follow-up (T3)
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). Change from baseline in the total WOMAC score (Likert scale version 3.1). The WOMAC assesses pain (5 items), stiffness (2 items), and physical function (17 items). Total score ranges from 0-96, with higher scores indicating worse symptoms/function.

SECONDARY OUTCOMES:
Change in Knee Range of Motion (Flexion and Extension) | Baseline (T0), Post-treatment (T2), 3-month Follow-up (T3)
  Change from baseline in active knee flexion and extension range of motion, measured in degrees using a standard goniometer.
Change in Functional Mobility | Baseline (T0), Post-treatment (T2), 3-month Follow-up (T3)
  Timed Up and Go Test (TUG). Change from baseline in the time (in seconds) taken to rise from a standard chair, walk 3 meters, turn, walk back, and sit down. Shorter times indicate better mobility.
Incidence of Adverse Events | Throughout study participation (up to 3-month follow-up)
  Number, type, and severity of any adverse events (AEs) reported by participants or observed by study staff throughout the study duration, particularly those potentially related to HILT (e.g., skin irritation, burns, increased pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Al Hayah University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No